CLINICAL TRIAL: NCT04780828
Title: Investigation of the Effects of Different Obesity Levels on the Respiratory System: In Our Study, Besides the Effect of Obesity on the Respiratory System, Many Different Parameters Related to Health Will be Compared.
Brief Title: Investigation of the Effects of Different Levels of Obesity on the Respiratory System
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Medipol University (Other)
Responsible Party: Principal Investigator, alihan bilen, physiotherapist, Istanbul Medipol University Hospital
Other Study IDs: 10840098-772.02-E.61593
Record Dates: First submitted 2021-02-23; First posted 2021-03-04 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Obesity, Adolescent; Obesity, Morbid; Obesity, Abdominal; Obesity, Visceral; Weight, Body
Keywords: Obesity; Respiratory System; Quality of Life; Anthropometric Measurements; Body Composition
MeSH Terms: conditions — Pediatric Obesity; Obesity, Morbid; Obesity, Abdominal; Body Weight; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- GROUP I: Group I will include cases classified as normal weight (healthy) with a body mass index of 18.5-24.9 kg / m2 as a result of the classification made by the World Health Organization. All parameter and evaluation measurements determined for this group will be made. Since this group was not considered as obese, it was determined as the control group.
- GROUP II: Group II will include cases classified as overweight and having a body mass index of 25.0-29.9 kg / m2 as a result of the classification made by the World Health Organization. All parameter and evaluation measurements determined in this group will be made.
- GROUP III: Group III will include cases classified as class I obese, with a body mass index of 30.0-34.9 kg / m2 as a result of the classification made by the World Health Organization. All parameter and evaluation measurements determined in this group will be made.
- GROUP IV: Group IV will include cases classified as class II obese, with a body mass index of 35.0-39.9 kg / m2 as a result of the classification made by the World Health Organization. All parameter and evaluation measurements determined in this group will be made.
- GROUP V: Group V will include cases classified as class III (morbid) obese, with a body mass index of 40 kg / m2 as a result of the classification made by the World Health Organization. All parameter and evaluation measurements determined in this group will be made.

SUMMARY:
Obesity can be defined as' a disease that occurs as a result of the energy (calorie) taken with food being more than the energy consumed and the excess energy being stored as fat in the body, negatively affecting the quality and duration of life. BMI is calculated by dividing the weight (kg) by the square of the height (m2) (1,2). According to the World Health Organization (WHO) classification, BMI between 25-29.9 kg / m2 is overweight, 30-34.9 kg / m2 is light, 35-39.9 kg / m2 is medium, 40 kg / m2 and above is considered as severe obesity. Obesity has important effects on respiratory function. These mechanical and biochemical effects are not easily measured by pulmonary function test and BMI measurement.Changes caused by mediators produced by adipose tissue likely cause changes in lung function, but this effect is not fully understood at the moment. The aim of our study is to make these effects more understandable and to compare them with different obesity classes and people with normal weight who are considered healthy.

Hypothesis 0: The effects of obesity on respiratory functions and multidimensional health-related parameters do not show a statistically significant difference compared to individuals with different levels of the disease and normal weight individuals classified as healthy.

Hypothesis 1: The effects of obesity on respiratory functions and multidimensional health-related parameters show a statistically significant difference compared to people with different levels of the disease and normal weight individuals classified as healthy.

The study will be carried out by face-to-face evaluations in a clinical setting with obese patients between the ages of 18-65 who have applied to the clinic with a diagnosis of obesity and agree to participate in the study, and healthy volunteers who are considered to be healthy without a diagnosis of obesity. Looking at the evaluations to be made; Measurement of respiratory function parameters, measurement of respiratory muscle strength, anthropometric measurements, evaluation of body composition, quality of life, upper extremity muscle strength and grip strength, lower extremity muscle strength, fatigue evaluation, vital signs, evaluation of exercise perception, presence of dyspnea and its level will be evaluated. A detailed description of these evaluations and the parameters to be used will be explained in detail in the next step.

DETAILED DESCRIPTION:
Obesity can be defined as' a disease that occurs as a result of the energy (calorie) taken with food being more than the energy consumed and the excess energy being stored as fat in the body, negatively affecting the quality and duration of life. A body mass index (BMI) of 30 or above in adults is classified as obese. BMI is calculated by dividing the weight (kg) by the square of the height (m2). According to the World Health Organization (WHO) classification, BMI between 25-29. 9 kg / m2 is overweight, 30-34. 9 kg / m2 is light, 35-39. 9 kg / m2 is medium, 40 kg / m2 and above is considered as severe obesity. As the increases in BMI are related to the number of comorbidities, weight loss also affects many risk factors. It has been shown that voluntary weight loss in obese individuals over short periods (weeks or months) reduces risk factors and improves disease symptoms associated with obesity, including heart disease, Type II Diabetes mellitus, and osteoarthritis. Obesity; It is an important risk factor and disease factor for asthma, obstructive sleep apnea syndrome, obesity hypoventilation syndrome (OHS) and pulmonary hypertension diseases. The overall effect of obesity on lung function is multifactorial and is related to the mechanical and inflammatory aspects of obesity. Obesity has important effects on respiratory function. These mechanical and biochemical effects are not easily measured by pulmonary function test and BMI measurement. Changes caused by mediators produced by adipose tissue likely cause changes in lung function, but this effect is not fully understood at the moment.As a result of the literature review the investigators conducted, it was observed that the studies conducted in order to make more understandable the physiological and mechanical effects of obesity on different systems in the body, especially the respiratory system, were limited and inadequate in terms of numerical and targeted purposes. It was observed that lower extremity muscle strength, fatigue, sleep quality parameters were not included, and their relations with respiratory system functions and measurements were not measured. The aim of our study is to make these effects more understandable and to compare them with different obesity classes and people with normal weight who are considered healthy. Individuals who volunteered to participate in the study, who met the inclusion criteria and volunteered to participate will be evaluated by dividing them into five different groups according to the BMI parameter, in accordance with the intervals determined by WHO, and the data obtained will be compared between the groups.

Outcome Measures:

* Measurement of Pulmonary Function Parameters: The respiratory function parameters of the participants will be measured with a respiratory function test using a spirometer. With these tests, the static and dynamic lung volumes and functional status of the person will be determined.
* Measurement of Respiratory Muscle Strength:

It consists of respiratory muscles, diaphragm, intercostal (internal and external), scalene, sternocleidomastoid, triangularis sterni, abdominal, shoulder and neck muscles. Respiratory muscle strength can be measured in many different ways. Among the pulmonary function tests, maximum inspiratory and expiratory pressures are the measurements that are frequently used to evaluate the strength of the respiratory muscles. -Measurement of Respiratory Muscle Strength:It consists of respiratory muscles, diaphragm, intercostal (internal and external), scalene, sternocleidomastoid, triangularis sterni, abdominal, shoulder and neck muscles. Respiratory muscle strength can be measured in many different ways. Among the pulmonary function tests, maximum inspiratory and expiratory pressures are the measurements that are frequently used to evaluate the strength of the respiratory muscles. These measurements are directly related to respiratory muscle strength and help to determine the rehabilitation and exercise program by providing information about the patient's condition.

-Anthropometric Measurements: Participants' waist circumference, hip circumference, neck circumference will be measured, and their ratios (waist / height ratio, waist / hip ratio) will be calculated. Body mass index (BMI), waist circumference, and waist-to-hip ratio (B / C) is the diagnostic methods commonly used to detect adiposity. Waist circumference and waist-hip ratio have been found to be useful measurements for measuring visceral fat accumulation. Measurement of neck circumference is used as an anthropometric marker to identify patients at risk for sleep apnea syndrome. At the same time, neck circumference is thought to be associated with other metabolic diseases. In addition to these measurements, the measurement called 'New BMI' used in the literature will also be made. In this measurement, BMI is calculated with the formula 1.3 × (kg / m2).

In order to calculate the body fat ratio, it is aimed to estimate the amount of body fat with the measurement of Clinica Universidad de Navarra-Body Adiposity Estimator (CUN-BAE) in addition to the bioelectric impedance method.

BMI measurement is insufficient to determine body fat and muscle ratio. Since it is difficult to determine the location of the fat tissue in the body, it will be evaluated with the '' Body Shape Index ''.

-Assessment of Body Composition: Body composition will be measured using the method called bioelectrical impedance analysis (BIA). This measurement is based on the principles of electrical conductivity of body tissues. It is a fast, practical and relatively inexpensive method compared to other similar devices and applications used to examine the body composition of individuals. This method shows the percentage and mass of body fat, lean body weight and the amount of water in the body and their distribution percentage. The person climbs on the device and places his or her hands in the designated places. Electric current travels through the body and provides information about parameters determined by certain algorithms and calculations.

-Quality of Life: Quality of life is accepted as a multidimensional structure with many different contents. Considering the decrease in physical capacity, pain, deterioration in interpersonal relationships, decreased self-esteem, loss of self-esteem, depression, social stigma, difficulty in finding a job, rejection by the school and business environment, it is understood how low the health-related quality of life of obese individuals is. In measuring the quality of life; Nottingham Health Profile questionnaire will be used. Nottingham Health Profile is a questionnaire consisting of 7 subtitles and 45 questions, including physical, social and psychological evaluations.

-Upper Extremity Muscle Strength and Gripping Strength: It is an important parameter related to muscle strength, functional capacity, cardiovascular disease risk factors and mortality. Upper extremity muscle strength and grip strength will be measured by hand dynamometer and weight lifting tests (arm curls test).

-Lower Extremity Muscle Strength: Abnormalities that usually occur in lower extremity muscles affect patients' physical performance and daily living activities, reduce exercise tolerance and impair health-related quality of life. 30-second sit-and-go test will be used to measure lower extremity muscle strength. The score is determined by the number of times the participant sits and stands up for 30 seconds from the moment the participant is commanded to place his hands on the crossed, shoulders in the chair he is sitting with his back supported and to start in the position where his feet are in full contact with the floor.

* Fatigue Assessment:

Fatigue is a common complaint in overweight and obese people. It has been stated that this is caused by increased body mass, decreased physical activity level and sleep disorders. In the assessment of fatigue, the Fatigue Severity Scale (39) will be used. The fatigue severity scale consists of 9 questions that question social relationship, physical performance and symptomatically the severity of fatigue. The total score is created according to the answers given to the questions.

-Vital Sign: Type 2 diabetes mellitus (T2DM), hypertension (HT), dyslipidemia (DLP), obstructive sleep apnea syndrome (OSAS) comorbidities have been associated with morbid obesity in obese individuals. Blood pressure, heart rate, oxygen saturation will be evaluated in order to observe the negative effects of these comorbidities.

-Evaluation of Exercise Perception: Aerobic exercise capacity is an essential component of physical fitness. Perceived benefits and perceived barriers to participating in physical activity will be assessed by Exercise Benefits / Barriers Scale (EBBS). It is a questionnaire consisting of 43 questions used to evaluate people's perception of exercise. Evaluates the ideas of being useful and preventive that exercise creates on people. The test score is determined by the score collected according to the answers given to the questions.

-Assessment of the Presence and Level of Dyspnea: According to the American Thoracic Society (ATS) report, the definition of dyspnea was defined as "unpleasant or uncomfortable breathing sensation and personal respiratory disturbance caused by various intensity senses" and it was stated to be a subjective feeling. "Modified Medical Research Council Scale (MMRC)" will be used to evaluate the presence of dyspnea. The MMRC is a five-item scale created on the basis of various activities that cause shortness of breath. The presence and effect of dyspnea occur according to the substance chosen by the person.

-Statistical method (s) to use: '' Hatem AM, Ismail MS, El-Hinnawy YH. 'Effect of different classes of obesity on the pulmonary functions among adult Egyptians: a cross-sectional study', Egypt J Bronchol 2019; 13: 510-5 '', the total number of samples determined for 5 groups in the sample size study, based on the FVC value and standard deviations in table 2, was calculated as 80 on the condition that it was 16 per group. Sample size calculation was made using the NCSS / PASS program. In the calculation, it was determined that the difference between the averages of the 5 groups should be 80% power and 95% confidence level to be significant. The statistical test method to be applied ANOVA will be used in conditions of normal distribution between groups, and Kruskal-Wallis test method will be used if the condition of normal distribution between groups cannot be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 18-65,
* body mass index ≥18.5 according to the World Health Organization (WHO) classification,
* Volunteering to participate in the study,

Exclusion Criteria:

* Accompanying neurological or orthopedic effects that will prevent participation in the study,
* Pregnancy status,
* Presence of a pacemaker,
* Having had Covid-19 disease ,
* Having had any thoracic or abdominal surgery or injury,
* For evaluation and control purposes Being unable to understand and apply the tests to be applied mentally and physically successfully,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: According to the WHO classification, the five groups to be formed will be group I normal weight (healthy), group II overweight, group III, class 1 obese, group IV, class 2 obese, group V, class 3 (morbid) obese.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Respiratory Function Parameters | Day 1.
  The respiratory function parameters of the participants will be measured with a pulmonary function test using a spirometer. With these tests, the static and dynamic lung volumes and functional status of the person will be determined. Spirometric measurements will be carried out by applying the guidelines for standardization of pulmonary function tests prepared by the American Thoracic Society (ATS) and the European Respiratory Society (ERS).

SECONDARY OUTCOMES:
Respiratory Muscle Strength | Day 1.
  Respiratory muscles are composed of diaphragm, intercostal (internal and external), scalene, sternocleidomastoid, triangularis sterni, abdominal, shoulder and neck muscles. Respiratory muscle strength can be measured in many different ways. The maximum inspiratory and expiratory pressures among the respiratory function tests are the measurements that are frequently used to evaluate the strength of the respiratory muscles. These measurements are directly related to respiratory muscle strengths and assist in determining the rehabilitation and exercise program by providing information about the patient's condition. Respiratory muscle strength measurements will be carried out in accordance with the standardization of the guidelines prepared by the American Thoracic Society (ATS) and the European Respiratory Society (ERS).
Measurement of Quality of Life | Day 1.
  Quality of life is accepted as a multidimensional structure with many different contents . In the measurement of quality of life; ''Nottingham Health Profile'' questionnaire will be used. Nottingham Health Profile is a questionnaire consisting of 7 subtitles and 45 questions including physical, social and psychological evaluations. This multifaceted scale includes: pain, emotional reactions, sleep, physical activity, energy and health status
Perception Of Exercise | Day 1.
  Aerobic exercise capacity is an essential component of physical fitness. Perceived benefits and perceived barriers to participating in physical activity will be assessed through the Exercise Benefits / Barriers Scale This scale consists of 43 multiple-choice questions. According to the answers given, the minimum score that can be taken is 43 and the maximum score is 172. The higher the score, the better the perception of people about exercise..

OTHER OUTCOMES:
Anthropometric Measurements Ratios | Day 1.
  Measuring the waist circumference, hip circumference and neck circumference and their ratios (waist / height ratio, waist / hip ratio) to each other will be calculated. Anthropometric measurements (height, weight, waist, neck and hip circumference) will be carried out according to the World Health Organization (WHO) measurement criteria. Measurements will be made with a 150 centimeter long tape measure that is not rigid.
Neck Circumference | Day 1.
  Measurement of neck circumference is used as an anthropometric marker to identify patients at risk for sleep apnea syndrome. Anthropometric measurements will be carried out according to the World Health Organization (WHO) measurement criteria. Measurements will be made with a 150 centimeter long tape measure that is not rigid.
Waist Circumference | Day 1.
  Waist circumference has been found to be useful measurements for measuring visceral fat accumulation. waist circumference is a frequently used diagnostic method for detecting adiposity. Waist circumference has been found to be useful measurements for measuring visceral fat accumulation. Anthropometric measurements will be carried out according to the World Health Organization (WHO) measurement criteria. Measurements will be made with a 150 centimeter long tape measure that is not rigid.
NEW BMI | Day 1.
  A measurement called 'New BMI' used in the literature will also be made. In this measurement, BMI is calculated with the formula 1.3 × (kg / m2).
Assessing Body Composition | Day 1.
  Body composition will be measured using the method called bioelectrical impedance analysis (BIA). With the device used in this method, the weight and height of the people are also measured. This measurement is based on the principles of electrical conductivity of body tissues. It is a fast, practical and relatively inexpensive method compared to other similar devices and applications used to examine the body composition of individuals. This method shows the percentage and mass of body fat, lean body weight and the amount of water in the body and their distribution percentage.
Body Adiposity Estimator | Day 1.
  In order to calculate the body fat ratio, it is aimed to estimate the amount of body fat with the measurement of Clinica Universidad de Navarra-Body Adiposity Estimator (CUN-BAE) in addition to the bioelectric impedance method. In this measurement,% BF (Percent estimate of body fat) = -44.988 (0.503 × age) (10.689 × gender) (3.172 × BMI) - (0.026 × BMI) (0.181 × BMI × gender) - (0.02 × BMI × age ) - (0.005 × BMI2 × gender) (0.00021 × BMI2 × age) (The multiplier value for the female gender is determined as 1, for the male gender the multiplier value is determined as 0)
Body Shape Index | Day 1.
  BMI measurement is insufficient to determine body fat and muscle ratio. Since it is difficult to determine the location of the fat tissue in the body, it will be evaluated with the "Body Shape Index" in this regard. Body Shape Index is calculated with the formula waist circumference (cm) / (BMI2 / 3 × Height (m) 1/2).
Body Adiposity Index | Day 1.
  Another parameter used to determine the body fat percentage is called the "Body Adiposity Index". A predictive value for the percentage of body fat is determined by the measurement result. Body Adiposity Index is calculated with the formula (hip circumference / Height (m) 1.5) -18.
Upper Extremity Muscle Strength | Day 1.
  In the weight lifting test to be used to measure upper extremity muscle strength, the score is determined by bringing the arm to full extension from the person (3.60 kg for male participants, 2.3 kg for female participants) and the number of full lifts for 30 seconds.In the weightlifting test to be used to measure upper extremity muscle strength, the score is determined by bringing the arm to full extension of the person (3.60 kg for male participants, 2.3 kg for female participants) and the number of full lifts for 30 seconds.
Gripping Strength | Day 1.
  Grip strength measurement is made using a hand dynamometer to measure the grip strength of the hand isometric.
Lower Extremity Muscle Strength | Day 1.
  Abnormalities that usually occur in lower extremity muscles affect patients' physical performance and activities of daily living, reduce exercise tolerance and impair health-related quality of life. 30-second sit-and-go test will be used to measure lower extremity muscle strength. The score is determined by the number of times the participant sits and stands up for 30 seconds from the moment the participant is commanded to place his hands on the crossed shoulders in the chair he is sitting with his back supported and to start in the position where his feet touch the floor.
Fatigue Assessment | Day 1.
  The fatigue severity scale consists of 9 questions that question social relationship, physical performance and symptomatically the severity of fatigue. The total score is created according to the answers given to the questions.The questions are scored between 0 and 7, and the result is obtained by dividing the total score by nine. As the total score increases, the severity of fatigue increases. If the result is less than 2.8, the result is found with no fatigue. If it is greater than 6.1, it is considered as chronic fatigue.
Blood Pressure | Day 1.
  Central adiposity has long been linked to hypertension in adults, with the finding that cardiovascular and metabolic complications of obesity were more common in patients with the upper body obesity phenotype. Blood pressure will be measured with a digital sphygmomanometer
Heart Rate | Day 1.
  Another important manifestation of obesity is impairment in the autonomic nervous system, present in all age groups, each of which has its own profile. Heart rate also changes due to this influence. Heart rate obtained using a heart rate monitor.
Oxygen Saturation | Day 1.
  Oxygen saturation is an important vital parameter. Oxygen saturation will be measured with a pulse oximeter.
Evaluation of the Presence and Level of Dyspnea | Day 1.
  According to the report of the American Thoracic Society (ATS), the definition of dyspnea was defined as "unpleasant or uncomfortable breathing sensation and personal respiratory distress caused by various intensity sensations '' and it was stated to be a subjective feeling. "Modified Medical Research Council Scale " will be used to evaluate the presence of dyspnea. The scale is a five-item scale based on various activities that cause shortness of breath. The presence and effect of dyspnea occurs according to the substance chosen by the person. In this scale consisting of five options, the effect created by the presence of dyspnea is determined according to the answer given. The lowest score is 0, the highest score is 5. Higher score means more exposure. And the higher the score, the worse the result.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Aras Bayram, Phd, Study Director — Medipol University
Locations (1):
- Istanbul University-Cerrahpaşa Faculty of Medicine Internal Medicine Department of Endocrinology and Metabolic Diseases, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of obesity in the United States, 2009-2010. NCHS Data Brief. 2012 Jan;(82):1-8. PMID 22617494
- [Background] Forhan M. An analysis of disability models and the application of the ICF to obesity. Disabil Rehabil. 2009;31(16):1382-8. doi: 10.1080/09638280802572981. PMID 19340616
- [Background] Sirtori A, Brunani A, Villa V, Berselli ME, Croci M, Leonardi M, Raggi A. Obesity is a marker of reduction in QoL and disability. ScientificWorldJournal. 2012;2012:167520. doi: 10.1100/2012/167520. Epub 2012 Mar 12. PMID 22536122
- [Background] Vranesic Bender D, Krznaric Z. Nutritional and behavioral modification therapies of obesity: facts and fiction. Dig Dis. 2012;30(2):163-7. doi: 10.1159/000336670. Epub 2012 Jun 20. PMID 22722432
- [Background] Bluher M. Obesity: global epidemiology and pathogenesis. Nat Rev Endocrinol. 2019 May;15(5):288-298. doi: 10.1038/s41574-019-0176-8. PMID 30814686
- [Background] The Lancet Public Health. Tackling obesity seriously: the time has come. Lancet Public Health. 2018 Apr;3(4):e153. doi: 10.1016/S2468-2667(18)30053-7. No abstract available. PMID 29627076
- [Background] Bray GA. Risks of obesity. Endocrinol Metab Clin North Am. 2003 Dec;32(4):787-804, viii. doi: 10.1016/s0889-8529(03)00067-7. PMID 14711062
- [Background] Laskowski ER. Action on obesity and fitness: the physiatrist's role. PM R. 2009 Sep;1(9):795-7. doi: 10.1016/j.pmrj.2009.08.448. No abstract available. PMID 19769911
- [Background] Raggi A, Sirtori A, Brunani A, Liuzzi A, Leonardi M. Use of the ICF to describe functioning and disability in obese patients. Disabil Rehabil. 2009;31 Suppl 1:S153-8. doi: 10.3109/09638280903317724. PMID 19968528
- [Background] Dixon AE, Peters U. The effect of obesity on lung function. Expert Rev Respir Med. 2018 Sep;12(9):755-767. doi: 10.1080/17476348.2018.1506331. Epub 2018 Aug 14. PMID 30056777
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] Wen AS, Woo MS, Keens TG. How many maneuvers are required to measure maximal inspiratory pressure accurately. Chest. 1997 Mar;111(3):802-7. doi: 10.1378/chest.111.3.802. PMID 9118723
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Chiu HY, Chen PY, Chuang LP, Chen NH, Tu YK, Hsieh YJ, Wang YC, Guilleminault C. Diagnostic accuracy of the Berlin questionnaire, STOP-BANG, STOP, and Epworth sleepiness scale in detecting obstructive sleep apnea: A bivariate meta-analysis. Sleep Med Rev. 2017 Dec;36:57-70. doi: 10.1016/j.smrv.2016.10.004. Epub 2016 Nov 5. PMID 27919588
- [Background] Onat A, Hergenc G, Yuksel H, Can G, Ayhan E, Kaya Z, Dursunoglu D. Neck circumference as a measure of central obesity: associations with metabolic syndrome and obstructive sleep apnea syndrome beyond waist circumference. Clin Nutr. 2009 Feb;28(1):46-51. doi: 10.1016/j.clnu.2008.10.006. Epub 2008 Nov 17. PMID 19010573
- [Background] Ahbab S, Ataoglu HE, Tuna M, Karasulu L, Cetin F, Temiz LU, Yenigun M. Neck circumference, metabolic syndrome and obstructive sleep apnea syndrome; evaluation of possible linkage. Med Sci Monit. 2013 Feb 13;19:111-7. doi: 10.12659/MSM.883776. PMID 23403781
- [Background] van Vugt JL, Cakir H, Kornmann VN, Doodeman HJ, Stoot JH, Boerma D, Houdijk AP, Hulsewe KW. The new Body Mass Index as a predictor of postoperative complications in elective colorectal cancer surgery. Clin Nutr. 2015 Aug;34(4):700-4. doi: 10.1016/j.clnu.2014.08.006. Epub 2014 Aug 15. PMID 25171837
- [Background] Gomez-Ambrosi J, Silva C, Catalan V, Rodriguez A, Galofre JC, Escalada J, Valenti V, Rotellar F, Romero S, Ramirez B, Salvador J, Fruhbeck G. Clinical usefulness of a new equation for estimating body fat. Diabetes Care. 2012 Feb;35(2):383-8. doi: 10.2337/dc11-1334. Epub 2011 Dec 16. PMID 22179957
- [Background] Bergman RN, Stefanovski D, Buchanan TA, Sumner AE, Reynolds JC, Sebring NG, Xiang AH, Watanabe RM. A better index of body adiposity. Obesity (Silver Spring). 2011 May;19(5):1083-9. doi: 10.1038/oby.2011.38. Epub 2011 Mar 3. PMID 21372804
- [Background] Krakauer NY, Krakauer JC. A new body shape index predicts mortality hazard independently of body mass index. PLoS One. 2012;7(7):e39504. doi: 10.1371/journal.pone.0039504. Epub 2012 Jul 18. PMID 22815707
- [Background] Faria SL, Faria OP, Cardeal MD, Ito MK. Validation study of multi-frequency bioelectrical impedance with dual-energy X-ray absorptiometry among obese patients. Obes Surg. 2014 Sep;24(9):1476-80. doi: 10.1007/s11695-014-1190-5. PMID 24464546
- [Background] Sarwer DB, Steffen KJ. Quality of Life, Body Image and Sexual Functioning in Bariatric Surgery Patients. Eur Eat Disord Rev. 2015 Nov;23(6):504-8. doi: 10.1002/erv.2412. PMID 26608946
- [Background] Niero M, Martin M, Finger T, Lucas R, Mear I, Wild D, Glauda L, Patrick DL. A new approach to multicultural item generation in the development of two obesity-specific measures: the Obesity and Weight Loss Quality of Life (OWLQOL) questionnaire and the Weight-Related Symptom Measure (WRSM). Clin Ther. 2002 Apr;24(4):690-700. doi: 10.1016/s0149-2918(02)85144-x. PMID 12017412
- [Background] Myers A, Rosen JC. Obesity stigmatization and coping: relation to mental health symptoms, body image, and self-esteem. Int J Obes Relat Metab Disord. 1999 Mar;23(3):221-30. doi: 10.1038/sj.ijo.0800765. PMID 10193866
- [Background] Kucukdeveci AA, McKenna SP, Kutlay S, Gursel Y, Whalley D, Arasil T. The development and psychometric assessment of the Turkish version of the Nottingham Health Profile. Int J Rehabil Res. 2000 Mar;23(1):31-8. doi: 10.1097/00004356-200023010-00004. PMID 10826123
- [Background] Oppert JM, Bellicha A, Roda C, Bouillot JL, Torcivia A, Clement K, Poitou C, Ciangura C. Resistance Training and Protein Supplementation Increase Strength After Bariatric Surgery: A Randomized Controlled Trial. Obesity (Silver Spring). 2018 Nov;26(11):1709-1720. doi: 10.1002/oby.22317. PMID 30358153
- [Background] Spruit MA, Sillen MJ, Groenen MT, Wouters EF, Franssen FM. New normative values for handgrip strength: results from the UK Biobank. J Am Med Dir Assoc. 2013 Oct;14(10):775.e5-11. doi: 10.1016/j.jamda.2013.06.013. Epub 2013 Aug 16. PMID 23958225
- [Background] Baillot A, Vallee CA, Mampuya WM, Dionne IJ, Comeau E, Meziat-Burdin A, Langlois MF. Effects of a Pre-surgery Supervised Exercise Training 1 Year After Bariatric Surgery: a Randomized Controlled Study. Obes Surg. 2018 Apr;28(4):955-962. doi: 10.1007/s11695-017-2943-8. PMID 28963710
- [Background] Maltais F, Decramer M, Casaburi R, Barreiro E, Burelle Y, Debigare R, Dekhuijzen PN, Franssen F, Gayan-Ramirez G, Gea J, Gosker HR, Gosselink R, Hayot M, Hussain SN, Janssens W, Polkey MI, Roca J, Saey D, Schols AM, Spruit MA, Steiner M, Taivassalo T, Troosters T, Vogiatzis I, Wagner PD; ATS/ERS Ad Hoc Committee on Limb Muscle Dysfunction in COPD. An official American Thoracic Society/European Respiratory Society statement: update on limb muscle dysfunction in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2014 May 1;189(9):e15-62. doi: 10.1164/rccm.201402-0373ST. PMID 24787074
- [Background] Bohannon RW, Crouch RH. Two-Minute Step Test of Exercise Capacity: Systematic Review of Procedures, Performance, and Clinimetric Properties. J Geriatr Phys Ther. 2019 Apr/Jun;42(2):105-112. doi: 10.1519/JPT.0000000000000164. PMID 29210933
- [Background] Mesarwi O, Polak J, Jun J, Polotsky VY. Sleep disorders and the development of insulin resistance and obesity. Endocrinol Metab Clin North Am. 2013 Sep;42(3):617-34. doi: 10.1016/j.ecl.2013.05.001. PMID 24011890
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Gils Contreras A, Bonada Sanjaume A, Montero Jaime M, Rabassa Soler A, Sabench Pereferrer F, Molina Lopez A, Becerra Tomas N, Del Castillo Dejardin D, Salas-Salvado J. Effects of Two Preoperatory Weight Loss Diets on Hepatic Volume, Metabolic Parameters, and Surgical Complications in Morbid Obese Bariatric Surgery Candidates: a Randomized Clinical Trial. Obes Surg. 2018 Dec;28(12):3756-3768. doi: 10.1007/s11695-018-3413-7. PMID 30109669
- [Background] Sechrist KR, Walker SN, Pender NJ. Development and psychometric evaluation of the exercise benefits/barriers scale. Res Nurs Health. 1987 Dec;10(6):357-65. doi: 10.1002/nur.4770100603. PMID 3423307
- [Background] FLETCHER CM. The clinical diagnosis of pulmonary emphysema; an experimental study. Proc R Soc Med. 1952 Sep;45(9):577-84. No abstract available. PMID 13003946
- [Background] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201
- See also: ''Waist Circumference and Waist to Hip Ratio: A Report of a WHO Expert Consultation'' — https://www.who.int/publications/i/item/9789241501491